CLINICAL TRIAL: NCT03278626
Title: A Phase I/II Open Label Multi Center Study of Immune Checkpoint Therapy With Nivolumab for Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Immune Checkpoint Therapy With Nivolumab Esophageal Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped earlier than anticipated due to slow accrual
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-00971
Record Dates: First submitted 2017-08-31; First posted 2017-09-11 (Actual); Results first posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Locally Advanced Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Nivolumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolimumab+Carboplatin/paclitaxel+Radiation (Other): 240 mg IVPB every 2 weeks for 2 doses, nivolumab at 240 mg every 2 weeks will be added to paclitaxel and carboplatin, which will be dosed according to the standard of care: paclitaxel 50 mg/m2 weekly for 6 weeks and carboplatin AUC 2 weekly for 6 weeks and radiation
  Interventions: Drug: Nivolimumab+Carboplatin/paclitaxel+Radiation

INTERVENTIONS:
Drug: Nivolimumab+Carboplatin/paclitaxel+Radiation — In the phase I portion of the study, up to six patients will be treated (radiation will be 50.4 Gy (1.8 Gy/fraction × 28 fractions)) and then observed for 28 days (following last day of treatment (Day 64)).
  Other Names: Opdivo; Paraplatin; Taxol

SUMMARY:
In this multi-institution phase I/II trial, the investigators have chosen paclitaxel and carboplatin using a schedule and doses identical to those used in the CROSS trial. Following a run-in with nivolumab alone at 240 mg IVPB every 2 weeks for 2 doses, nivolumab at 240 mg every 2 weeks will be added to paclitaxel and carboplatin, which will be dosed according to the standard of care established by the CROSS trial: paclitaxel 50 mg/m2 weekly for 6 weeks and carboplatin AUC 2 weekly for 6 weeks. Concurrent radiation will be administered with chemotherapy at 1.8 Gy/fraction × 28 fractions to a total dose of 50.4 Gy, the standard radiation dose administered in the United States for trimodality therapy that includes concurrent therapy with carboplatin and paclitaxel. A decrease in dose to 41.4 Gy per the protocol established by van Hagen, et al. will be permitted before discontinuing therapy due to unacceptable toxicity. While the CROSS study administered only 5 weekly doses of chemotherapy during the 5 weeks of radiation, the higher dose of 50.4 Gy (1.8 Gy/fraction ×28 fractions over 5½ weeks) utilized in this study permits for a sixth dose during the additional week of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, treatment-naive esophageal squamous cell carcinoma
* Previously obtained archival tumor tissue, or tissue obtained by endoscopically guided core biopsy at screening
* TanyN1-3 or T3-4 N0as determined by EUS and PET/CT. All palpable or CT/PET visible lymph nodes outside the usual surgical field must be biopsy-proven negative for cancer.
* All patients must have locoregional staging determined by endoscopic ultrasound (EUS) if technically feasible. Endoscopy reports or subsequent GI clinic note should clearly state both the T and N stage.
* All patients must have initial PET/CT scans to document no evidence of metastatic or unresectable squamous cell cancer
* All patients with tumors involving the thoracic esophagus must undergo bronchoscopy to document the absence of a fistula No known contraindication to the use of taxanes or platinum compounds.
* No history of severe hypersensitivity reaction to Cremophor® EL.
* Patients who are ≥ 18 years old are eligible for this study. Neither specific gender distribution, nor specific racial or ethnic origins are necessary for enrollment in this study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* A patient must be capable of giving informed consent or have an acceptable surrogate capable of giving consent on the subject's behalf
* Deemed a suitable candidate for esophagectomy by the treating surgeon as documented in a pre-operative assessment visit per standard practice at each participating institution.
* Deemed a suitable candidate for radiation therapy by the treating radiation oncologist as documented in a standard pretreatment visit per standard practice at each participating institution.
* Patient must be non-pregnant and non-nursing. Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to C1D1.
* Screening Laboratory Values must meet the following criteria and should be obtained within 14 days prior to C1D1 (see Table 1 below)
* Patients with a positive Hepatitis B core antibody (HBVcAb) must have negative viral load measurement; Patients with HBV core positive, must have negative viral load measurements
* Screening Laboratory Values must meet the following criteria and should be obtained within 14 days prior to randomization/registration (see Table 1 below) Test Acceptable Result WBC ≥ 2000/µL Neutrophils ≥ 1500/µL Platelets ≥ 100,000 /µL Hemoglobin > 9.0 g/dL Serum Creatinine ≤ 1.5 x ULN OR Creatinine Clearance (CrCl)* ≥ 40 mL/min AST ≤ 3 x ULN ALT ≤ 3 x ULN Total Bilirubin** ≤ 1.5 x ULN

Oxygen Saturation (O2 Sat.) ≥92% on ambient air Hepatitis B status HBV Surface Antigen Negative HBV Surface Antibody Positive or Negative HBV Core Antibody Negative Hepatitis C status Anti-HCV Total Antibody Negative HCV RNA analysis Negative HIV status Rapid HIV 1/2 Antibodies Negative *Creatinine Clearance Calculated using the Cockcroft-Gault formula

Female CrCl = (140- age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL

Male CrCl = (140- age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL

**Total Bilirubin ≤ 1.5 x ULN, except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL

Exclusion Criteria:

* T1-2 N0 as determined by EUS and PET/CT.
* Pregnant or lactating women
* Active or prior documented autoimmune or inflammatory disorders including but not limited to inflammatory bowel disease; systemic lupus erythematosus; type I diabetes mellitus; Wegener syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis, hypophysitis, uveitis) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:
* Subjects with vitiligo or alopecia
* Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest Computed Tomography (CT) scan
* The use of immunosuppressive medication within 28 days prior to the first dose of nivolumab. The following are exceptions to this criterion:
* Intranasal, topical, inhaled corticosteroids or local steroid injections (e.g. intra-articular injection)
* Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent
* Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication
* Positive test for Human Immunodeficiency Virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Active Hepatitis B or Hepatitis C (defined as positive-HBV surface antigen or detectable HCV-antibody) indicating acute or chronic infection. Patients with a positive Hepatitis B core antibody (HBVcAb) must have negative viral load measurement.
* Prior treatment with any immunotherapy
* Any other factors, including psychiatric or social, that in the opinion of the treating physician makes the patient an inappropriate candidate for a study.
* Patients are excluded if they have active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for [lowest minimum is 4 weeks or more] after treatment is complete and within 28 days prior to the first dose of nivolumab administration. There must also be no ESCC Nivolumab requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* As there is potential for hepatic toxicity with nivolumab or nivolumab non-drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Patients with a history of allergy to the study drug components are excluded.
* No herbal supplements are allowed in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wu, MD, Principal Investigator — NYU Langone Health
Locations (5):
- United States (5):
  - University of Califonia, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - New York University School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health Sciences University, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolimumab+Carboplatin/Paclitaxel+Radiation
Started | 12
Completed | 7
Not Completed | 5
Not completed — Death | 2
Not completed — Toxicity | 1
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Population: 6 subjects enrolled in Phase 1, and 6 subjects enrolled in Phase 2
Arm/Group | Nivolimumab+Carboplatin/Paclitaxel+Radiation
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 63.95 [47.03 to 86.17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Unacceptable Toxicity (UT) Events
Description: UT is defined as:
  1. Recurrent grade 3 or 4 hematologic toxicity (despite 1 prior dose reduction in chemotherapy)
  2. any toxicity that results in a > 2-week delay in chemoradiation
Time Frame: 92 days (up to 28 days after Day 64)
Measure: Number; unit: Unacceptable Toxicity Events
Arm/Group | Nivolimumab+Carboplatin/Paclitaxel+Radiation
Number analyzed (Participants) | 6
Unacceptable Toxicity Events | 0

2. Primary Outcome: Phase 2: Number of Subjects Who Achieved cCR (Clinical Complete Response) or pCR (Pathological Complete Response)
Description: Clinical and pathological response after neoadjuvant therapy cCR by endoscopic + PET/CT evaluation; pCR for patients undergoing surgery Clinical Complete Response (cCR), no malignancy is found on clinical examination, imaging, endoscopy, and biopsy; Pathological Complete Response (pCR), no invasive and no in situ residual tumors in tissue
Time Frame: 5-8 Weeks post radiation treatment (7-8 months after treatment start)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolimumab+Carboplatin/Paclitaxel+Radiation
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: 100 days post-treatment
Arm/Group | Nivolimumab+Carboplatin/Paclitaxel+Radiation
All-Cause Mortality (participants affected / at risk) | 2/12
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolimumab+Carboplatin/Paclitaxel+Radiation (N=12)
Abdominal Pain (Gastrointestinal disorders) | 1
Lung Infection (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Fever (General disorders) | 1
Confusion (Psychiatric disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Rash-Morbiliform (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolimumab+Carboplatin/Paclitaxel+Radiation (N=12)
Abdominal Pain (Gastrointestinal disorders) | 3
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthralgia Knee Pain (Musculoskeletal and connective tissue disorders) | 1
Aspartate Aminotransferase Increased (Investigations) | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 5
Ataxia (Nervous system disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Chest Pain After Stent (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Decreased Lymphocyte Count (Investigations) | 10
Decreased Neutrophil Count (Investigations) | 7
Decreased Platelet Count (Investigations) | 9
Decreased Wbc Count (Investigations) | 9
Dehydration (Metabolism and nutrition disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis Radiation (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 8
Dyspnea (Gastrointestinal disorders) | 3
Esophageal Discomfort (Gastrointestinal disorders) | 1
Esophageal Pain (Gastrointestinal disorders) | 5
Esophagitis (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 6
Fever (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 6
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (General disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 2
Increased Blood Bilirubin (Investigations) | 4
Increased Wbc (Investigations) | 1
Infusion Related Reaction (General disorders) | 1
INR Increased (Investigations) | 2
Intermittent Non Cardiac Chest Pain (General disorders) | 1
Left Hip Pain (Musculoskeletal and connective tissue disorders) | 1
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1
Low Tsh (Investigations) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Night Sweats (General disorders) | 1
Nose Bleed (General disorders) | 1
Odynophagia (General disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Post Operation Pain (General disorders) | 1
Presyncope (Nervous system disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4
Rash-Morbiliform (Skin and subcutaneous tissue disorders) | 4
Rectal Bleeding (General disorders) | 1
Syncope (Nervous system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Upper Back Pain (Musculoskeletal and connective tissue disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 4
Vomiting After Stent (Gastrointestinal disorders) | 1
Weight Loss (Investigations) | 3
Alt Increased (Investigations) | 3
Ast Increased (Investigations) | 3
Increased Alk Phos (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03278626/Prot_SAP_000.pdf